CLINICAL TRIAL: NCT01198886
Title: Vitality, Independence, and Vigor in Elders Study (VIVE Study): Effects of an Exercise and Nutrition Program on Functionality in the Elderly
Brief Title: The Vitality, Independence, and Vigor in Elders Study I Clinical Trial
Acronym: VIVE-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 1006010; 09.37.CLI (Other Grant/Funding Number: Nestle Nutrition)
Record Dates: First submitted 2010-09-08; First posted 2010-09-10 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Functionally Limited; Sedentary
Keywords: Mobility disability; Older adults; Physical activity; Nutritional status
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Successful Aging Program (Placebo Comparator)
  Interventions: Other: Successful Aging Program
- Exercise-Nutrition Program (Experimental)
  Interventions: Other: Exercise-Nutrition Program

INTERVENTIONS:
Other: Successful Aging Program — Once per week discussion on lifestyle topics important to older adults. Classes conclude with a gentle upper body stretching routine.
  Arms: Successful Aging Program
Other: Exercise-Nutrition Program — Targeted exercise program offered 3-days per week at the study participants place of residence (senior housing facility). Other means to encourage physical activity outside of these exercise classes will be available. A nutrient-rich protein carbohydrate experimental beverage will be taken following the exercise sessions.
  Arms: Exercise-Nutrition Program

SUMMARY:
The primary objective of this study is to evaluate changes in functional status that result from an Exercise-Nutrition Program (ENP) targeted toward older adults residing at senior housing facilities.

- The primary hypothesis is that over the 6-month intervention period subjects in the intervention group will realize significant improvements in lower extremity function compared to a control group.

Secondary objectives

To evaluate changes in nutritional status that result from the ENP.

- The secondary hypothesis is that subjects in the intervention group will realize significant increases in circulating insulin-like growth factor-1 (IGF-1) and 25-hydroxy vitamin D (25(OH)D) and demonstrate improvements in nutritional status compared to a control group.

To evaluate changes in inflammatory status that result from the ENP.

- Subjects in the ENP group will exhibit reduced concentrations of circulating interleukin-6 (IL-6) compared with the control group.

To evaluate changes in psychosocial factors that result from the ENP

* The related hypothesis is that over the 6-month intervention period subjects in the intervention group will increase exercise self-efficacy, intrinsic motivation to exercise, and satisfaction of psychological needs compared to a control group.
* Additionally it is hypothesized that subjects in the intervention group will realize improvements in mood and quality of life compared to a control group.

To assess the feasibility of conducting the Exercise-Nutrition Program in a senior housing facility setting.

DETAILED DESCRIPTION:
Older adults are the fastest growing segment of the population in many countries around the world, and the maintenance of independence has emerged as a major public health priority. Although a significant decline in physical function was once considered an inevitable consequence of aging, many studies have demonstrated that targeted exercise programs can dramatically improve physical function, even into advanced age. There is also evidence that appropriately timed protein intake is important for exercise recovery and the growth and maintenance of lean body mass. Other nutrients may be important to muscle strength and function as well. Yet many older adults have poor nutritional status. A combined exercise and nutrition program for functionally at-risk older adults, conveniently offered in the senior housing facilities where many reside, has great potential to improve functional status and quality of life in this population.

Main objective

* The primary objective of this study is to evaluate changes in functional status that result from the Exercise-Nutrition Program (ENP).
* The primary hypothesis is that over the 6-month intervention period subjects in the intervention group will realize significant improvements in lower extremity function compared to a control group.

Secondary objectives

The secondary objectives of the research project are:

* To evaluate changes in nutritional status that result from the ENP.
* The secondary hypothesis is that subjects in the intervention group will realize significant increases in circulating IGF-1 and 25-hydroxy vitamin D (25(OH)D) and demonstrate improvements in nutritional status compared to the control group.
* Subjects in the ENP will exhibit reductions in circulating plasma IL-6 concentrations, which are indicative of systemic inflammatory status.
* To evaluate changes in psychosocial factors that result from the ENP.
* The related hypothesis is that over the 6-month intervention period subjects in the intervention group will increase exercise self-efficacy, intrinsic motivation to exercise, and satisfaction of psychological needs compared to a control group.
* Additionally it is hypothesized that subjects in the intervention group will realize improvements in mood and quality of life compared to a control group.

Another major objective is to assess the feasibility of conducting the Exercise-Nutrition Program in a senior housing center facility setting.

TRIAL DESIGN

Type of trial The study objectives will be achieved in the context of a controlled, randomized field trial. Randomization will be by site (senior housing center). Intervention group subjects will participate in the Exercise-Nutrition Program (ENP). Control group subjects will participate in the Successful Aging Program (SAP), which will provide them with useful skills and an adequate attention control, but will not affect the primary outcome of this study.

Subjects, groups and centers:

In each study group the number of subjects to complete the study protocol will be 40 (see also 9.3 statistical section). Assuming a conservative dropout rate of 10% after the 3 month intervention and 15% at the end of the 6 month study, a sample of 53 subjects per group, or 106 total, will be required to be enrolled in the study. 16-20- senior housing centers will be recruited and each will run one class with an average size of at least 5 subjects (maximum 25 subjects).

Sites will be assigned to one of 2 groups:

Group 1: Exercise-Nutrition Program (ENP) Group 2: Successful Aging Program (SAP)

Duration of subject participation:

Subjects will undergo the proposed intervention for 6 months. The target population for this study will be elderly people (65 yrs+) living in senior housing centers.

ELIGIBILITY:
Inclusion Criteria:

* Age 65+
* Living at a senior housing facility
* SPPB score of 3-9
* BMI <35
* 6CIT < or = 14
* Permission of primary care provider
* Willingness to be randomized to either treatment group

Exclusion Criteria:

* Failure to provide informed consent
* Participate in >125 minutes per week of moderate to vigorous physical activity
* Moderate to severe cognitive impairment (6CIT >15)
* Inability to communicate due to severe, uncorrectable hearing loss or speech disorder
* Severe visual impairment (if it precludes completion of assessments and/or intervention)
* Wheelchair bound
* Late-stage, progressive, degenerative neurologic disease, e.g., Parkinson's Disease, multiple sclerosis, acute lateral sclerosis.
* Severe rheumatologic or orthopedic diseases, e.g., awaiting joint replacement, active inflammatory disease
* Terminal illness with life expectancy less than 12 months, as determined by a physician
* Severe pulmonary disease, requiring either steroid pills or injections or the use of supplemental oxygen
* Severe cardiac disease, including NYHA Class III or IV congestive heart failure, clinically significant aortic stenosis, history of cardiac arrest, use of a cardiac defibrillator, or uncontrolled angina
* Other significant co-morbid disease that would impair ability to participate in the exercise-based intervention, e.g. renal failure on hemodialysis, severe psychiatric disorder (e.g. bipolar, schizophrenia), excessive alcohol use (>14 drinks per wk); persons with depression will not be excluded
* Surgery in the previous 6 months
* Patient who cannot be expected to comply with treatment
* Inability to obtain signed authorization from participant's primary care health care provider.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 121 (Actual)
Dates: Start 2010-09; Primary Completion 2013-01 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Short Physical Performance Battery (SPPB) | Baseline, 3 months, 6 months, and 12 months into the study
  Tests of functional mobility that include strength and balance. Appropriate for older adults.

CONTACTS AND LOCATIONS:
Overall Officials: Miriam E Nelson, PhD, Study Director — Tufts University; Sara C. Folta, PhD, Principal Investigator — Tufts University; Roger F. Fielding, PhD, Principal Investigator — Tufts University
Locations (17):
- United States (17):
  - Drake Village, Arlington, Massachusetts
  - Nashoba Park, Ayer, Massachusetts
  - Compass on the Bay, Boston, Massachusetts
  - Chestnut Park at Cleveland Circle, Brighton, Massachusetts
  - Neville Place at Fresh Pond, Cambridge, Massachusetts
  - Youville House, Cambridge, Massachusetts
  - Chelmsford Crossings, Chelmsford, Massachusetts
  - Putnam Farms at Danvers, Danvers, Massachusetts
  - Standish Village at Lower Mills, Dorchester, Massachusetts
  - Youville Place, Lexington, Massachusetts
  - Methuen Village, Methuen, Massachusetts
  - Evans Park at Newton Center, Newton, Massachusetts
  - Coleman House, Newton, Massachusetts
  - The Falls at Cordingly Dam, Newton, Massachusetts
  - Golda Meir House, Newton, Massachusetts
  - Holland Street Center, Somerville, Massachusetts
  - Waltham Crossings, Waltham, Massachusetts

REFERENCES:
- [Derived] Corcoran MP, Chui KK, White DK, Reid KF, Kirn D, Nelson ME, Sacheck JM, Folta SC, Fielding RA. Accelerometer Assessment of Physical Activity and Its Association with Physical Function in Older Adults Residing at Assisted Care Facilities. J Nutr Health Aging. 2016;20(7):752-8. doi: 10.1007/s12603-015-0640-7. PMID 27499309